CLINICAL TRIAL: NCT00878722
Title: A Phase I/II Clinical Trial of PXD101 in Combination With Idarubicin in Patients With AML Not Suitable for Standard Intensive Therapy
Brief Title: Trial of PXD101 (Belinostat) in Combination With Idarubicin to Treat AML Not Suitable for Standard Intensive Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PXD101-CLN-15
Record Dates: First submitted 2009-04-07; First posted 2009-04-09 (Estimated); Results first posted 2014-11-13 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; PXD101; Belinostat; Idarubicin
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — belinostat; Idarubicin

ARMS (2):
- Arm A (Experimental): PXD101 administered as a 30-minute intravenous (IV) infusion of 1000 mg/m²/d for five consecutive days every 3 weeks.
  Idarubicin administered on day 5 (first steps) or days 4 and 5 (later steps). Patients will be treated in a 21-day cycle for a minimum of 2 cycles and a maximum of 6 cycles (depending on cumulated idarubicin dose).
  Interventions: Drug: PXD101; Drug: idarubicin
- Arm B (Experimental): PXD101 administered by continuous intravenous infusion over 24-48 hours and idarubicin (in the later steps) added after the first 24 hours. The second cycle will start on day 15 but under observation of possible toxicity. Further cycles will be administered q 14 d for up to 6 cycles. The first dose steps will be carried out with PXD101 alone for safety reasons.
  Interventions: Drug: PXD101; Drug: idarubicin

INTERVENTIONS:
Drug: PXD101
  Other Names: Belinostat
Drug: idarubicin
  Other Names: Zavedos

SUMMARY:
An open-label, non-randomized, multi-centre, Phase I/II trial to assess the efficacy and safety of 2 schedules of PXD101 in combination with idarubicin in patients with AML not suitable for standard intensive therapy.

DETAILED DESCRIPTION:
This trial is an open-label, multi-centre, dose-escalation Phase I/II study to evaluate safety, explore efficacy, pharmacodynamics, and pharmacokinetics of the combination of PXD101 with idarubicin administered in two different schedules in patients with AML. The PXD101 plus idarubicin treatment will be repeated at suitable intervals (target is every 3 weeks for schedule A and every 2 weeks for schedule B) depending upon toxicities or disease progression. Safety and efficacy assessments will be performed at every cycle.

Schedule A uses PXD101 by 30 min infusion daily for 5 days every 3 weeks with escalating doses of idarubicin.

Schedule B uses escalating doses of continuous infusion (48h) of PXD101 alone or in combination with idarubicin.

In both regimens the trial may be expanded at the Maximum Tolerated Dose (MTD).

ELIGIBILITY:
Inclusion Criteria: (abbreviated)

1. Signed consent
2. AML patients:

   1. above 60 years in first relapse or refractory.
   2. 18-60 years 2nd relapse or refractory to at least two intensive chemotherapy regimens.
   3. above 60 years with high risk features (cytogenetics, secondary or treatment related AML) d) above 60 years with myelodysplastic syndrome with >10% blasts in bone marrow (WHO RAEB-2 (Refractory anemia with excess blasts-2)). For patients below 60 years potential curative treatments should have been exhausted.
3. Performance status (ECOG) ≤ 2
4. Age ≥ 18 years
5. Acceptable liver, renal and bone marrow function as defined
6. Serum potassium within normal range.
7. Acceptable coagulation status as defined
8. Precautions for female patients with reproductive potential as defined

Exclusion Criteria:

1. Treatment with investigational agents within the last 4 weeks
2. Prior treatment with HDAC (Histone deacetylases) inhibitors including valproic acid
3. Prior anti-leukemic therapy (except hydroxyurea) within the last 3 weeks of trial dosing
4. Co-existing active infection (including HIV) or any co-existing medical condition likely to interfere with trial procedures, including significant cardiovascular disease
5. Altered mental status precluding understanding of the informed consent process and/or completion of the necessary study procedures.
6. Concurrent second malignancy.
7. History of hypersensitivity to idarubicin
8. Cumulative idarubicin dose exceeding 100 mg/m², or a (with respect cardiotoxicity) corresponding dose of other anthracyclines
9. LVEF (left ventricular ejection fraction) below normal range (< 45% )
10. Known Central Nervous System (CNS) leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-08; Primary Completion 2009-05 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: e-mail contact via enquiries@topotarget.com, Study Chair — Valerio Therapeutics
Locations (6):
- France (2):
  - CHU Lapeyronie, Montpellier
  - Hôpital St. Louis, Paris
- Germany (3):
  - Uniklinik Homburg, Homburg
  - Uni Hospital Marburg, Marburg
  - Universitätsklinikum Ulm, Ulm
- Christie Hospital NHS Trust, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A, Step 1: PXD101 (belinostat) 1000 mg/m²/d for 5 consecutive days every 3 weeks. On day 5, Idarubicin 5 mg/m²
- Arm A, Step 2: PXD101 1000 mg/m²/d for 5 consecutive days every 3 weeks. On day 5, Idarubicin 10 mg/m²
- Arm A, Step 3: PXD101 1000 mg/m²/d for 5 consecutive days every 3 weeks. On days 4 and 5, Idarubicin 7.5 mg/m²/d
- Arm A, Step 4: PXD101 1000 mg/m²/d for 5 consecutive days every 3 weeks. On days 4 and 5, Idarubicin 10 mg/m²/d
- Arm B, Steps 1-6: PXD101 administered by continuous intravenous infusion over 24-48 hours, doses 25 mg/m²/24 hours to 800 mg/m²/24 hours for 48 hours
- Arm B, Step 7: PXD101 administered by continuous intravenous infusion over 48 hours, dose 1000 mg/m²/48 hours
  Idarubicin added at 5 mg/m² after 48 hours. Further cycles will be administered q 14 d for up to 6 cycles
- Arm B, Step 8: PXD101 administered by continuous intravenous infusion over 48 hours, dose 1000 mg/m²/48 hours
  Idarubicin added at 5 mg/m² after 24 and 48 hours. Further cycles will be administered q 14 d for up to 6 cycles
- Arm B, Step 9: PXD101 administered by continuous intravenous infusion over 48 hours, dose 1000 mg/m²/48 hours
  Idarubicin added at 7.5 mg/m² after 24 and 48 hours. Further cycles will be administered q 14 d for up to 6 cycles
Period: Overall Study
Arm/Group | Arm A, Step 1 | Arm A, Step 2 | Arm A, Step 3 | Arm A, Step 4 | Arm B, Steps 1-6 | Arm B, Step 7 | Arm B, Step 8 | Arm B, Step 9
Started | 3 | 3 | 3 | 9 | 7 | 3 | 6 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 3 | 3 | 3 | 9 | 7 | 2 | 6 | 7
Not completed — Progressive disease | 3 | 3 | 3 | 7 | 7 | 1 | 4 | 3
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Relapse | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A, Step 1: PXD101 1000 mg/m²/d for 5 consecutive days every 3 weeks. On day 5, Idarubicin 5 mg/m²
- Total: Total of all reporting groups
Arm/Group | Arm A, Step 1 | Arm A, Step 2 | Arm A, Step 3 | Arm A, Step 4 | Arm B, Steps 1-6 | Arm B, Step 7 | Arm B, Step 8 | Arm B, Step 9 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9 | 7 | 3 | 6 | 7 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 3 | 4 | 0 | 3 | 3 | 16
  >=65 years | 2 | 2 | 2 | 6 | 3 | 3 | 3 | 4 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 0 | 1 | 4 | 1 | 5 | 2 | 16
  Male | 3 | 0 | 3 | 8 | 3 | 2 | 1 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose, Dose Limiting Toxicity
Description: DLT (dose limiting toxicities): patients with any of the toxicities: 1.Haematological toxicity is not included in the definition due to bone marrow involvement by the disease except for following grade 4 ANC (absolute neutrophil count) and PLT (platelet count) for 6 weeks with less than 5% blasts in bone marrow. 2.Drug related non hematological Grade 3 or 4 toxicity except alopecia, brief nausea and vomiting, diarrhea, rash, arthralgias and myalgias. Treatment interventions should palliate toxicity symptoms prior to concluding a DLT has occurred (e.g if nausea and vomiting to Grade 3 have been associated with the drug). If despite standard treatment Grade 3 nausea and or vomiting persisted then a DLT was considered to have occurred. Grade 4 diarrhea in spite of standard therapeutic measures was included in DLT definition. 3.Inability to tolerate full dosing cycle due to toxicity or any drug-related adverse event resulting in more than 14 day treatment delay in the next treatment cycle
Time Frame: First Cycle
Measure: Number; unit: participants
Arm/Group | Arm A, Step 1 | Arm A, Step 2 | Arm A, Step 3 | Arm A, Step 4 | Arm B, Steps 1-6 | Arm B, Step 7 | Arm B, Step 8 | Arm B, Step 9
Number analyzed (Participants) | 3 | 3 | 3 | 9 | 7 | 3 | 6 | 7
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Overall Response
Description: Efficacy measured as Response rate (complete response ([CR] and Complete remission with incomplete recovery of platelets [CRi]) and partial response ([PR])) using the response criteria of the International Working Group (Cheson et al 2003). CR includes CRi, CRc (Cytogenetic complete remission), and CRm (Molecular complete remission).
Time Frame: Throughout study, after each cycle for the first two cycles, then after every second cycle
Measure: Number; unit: participants
Arm/Group | Arm A, Step 1 | Arm A, Step 2 | Arm A, Step 3 | Arm A, Step 4 | Arm B, Steps 1-6 | Arm B, Step 7 | Arm B, Step 8 | Arm B, Step 9
Number analyzed (Participants) | 3 | 3 | 3 | 9 | 7 | 3 | 6 | 7
participants | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 3

3. Secondary Outcome: Time to Response (CR and PR)
Description: Time to response: time in weeks from first treatment to obtainment of the particular response status (CR and PR)
Time Frame: Throughout study, after each cycle for the first two cycles, then after every second cycle
Population: Time to response was reported among participants who reported response
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Arm A, Step 1 | Arm A, Step 2 | Arm A, Step 3 | Arm A, Step 4 | Arm B, Steps 1-6 | Arm B, Step 7 | Arm B, Step 8 | Arm B, Step 9
Number analyzed (Participants) | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 3
Weeks |  | 2.6 [NA to NA] — Only 1 patient analyzed | 7.9 [NA to NA] — Only 1 patient analyzed | 6.0 [NA to NA] — Only 1 patient analyzed | 4.0 [NA to NA] — Only 1 patient analyzed | 1.9 [NA to NA] — Only 1 patient analyzed | 4.0 [NA to NA] — Only 1 patient analyzed | 1.0 [0.6 to 2.1]

4. Secondary Outcome: Duration of Response (CR and PR)
Description: Duration of Response (CR and PR) in Weeks
Time Frame: Throughout study, after each cycle for the first two cycles, then after every second cycle
Population: All patients who received at least one dose of belinostat and/or idarubicin were included in the full analysis set (FAS). Duration of response was reported among participants who reported response
Measure: Mean (Full Range); unit: weeks
Arm/Group | Arm A, Step 1 | Arm A, Step 2 | Arm A, Step 3 | Arm A, Step 4 | Arm B, Steps 1-6 | Arm B, Step 7 | Arm B, Step 8 | Arm B, Step 9
Number analyzed (Participants) | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 3
weeks |  | 26.3 | 20.6 | 28.1 | 5.4 | 30.3 | 19.6 | 4.3 [3 to 6.1]

5. Secondary Outcome: Overall Survival
Description: Overall survival: time in weeks from entry into study until death from any cause. All patients without this endpoint at the time of discontinuation or the end of trial have been censored.
Time Frame: Throughout study, after each cycle for the first two cycles, then after every second cycle
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Arm A, Step 1 | Arm A, Step 2 | Arm A, Step 3 | Arm A, Step 4 | Arm B, Steps 1-6 | Arm B, Step 7 | Arm B, Step 8 | Arm B, Step 9
Number analyzed (Participants) | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 3
Weeks |  |  |  | 10 [3.0 to 10.3] | 4.9 [2.0 to 7.9] | 3.7 [3.7 to 3.7] |  | 3.9 [0.7 to 9.9]

6. Secondary Outcome: Relapse-Free Survival
Description: Relapse-free survival: time (weeks) from leukemia-free state to relapse or death from any cause.
Time Frame: Throughout study, after each cycle for the first two cycles, then after every second cycle
Population: Relapse free survival was reported among participants who reported response
Measure: Number; unit: Weeks
Arm/Group | Arm A, Step 1 | Arm A, Step 2 | Arm A, Step 3 | Arm A, Step 4 | Arm B, Steps 1-6 | Arm B, Step 7 | Arm B, Step 8 | Arm B, Step 9
Number analyzed (Participants) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1
Weeks |  | 26.3 | 20.6 | 28.1 |  | 30.3 |  | 6.1

7. Secondary Outcome: Event-Free Survival
Description: Event-free survival: time (weeks) from entry into study until treatment failure, disease relapse or death from any cause.
Time Frame: Throughout study, after each cycle for the first two cycles, then after every second cycle
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Arm A, Step 1 | Arm A, Step 2 | Arm A, Step 3 | Arm A, Step 4 | Arm B, Steps 1-6 | Arm B, Step 7 | Arm B, Step 8 | Arm B, Step 9
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 7 | 3 | 5 | 5
Weeks | 5.1 [2.1 to 10.9] | 3.1 [1.9 to 28.7] | 8.0 [6.7 to 28.3] | 6.5 [3.0 to 10.3] | 2.0 [0.4 to 7.9] | 5.4 [3.4 to 32.1] | 5.4 [4.1 to 26.0] | 6.4 [0.7 to 9.9]

8. Secondary Outcome: Remission Duration
Description: Remission duration: time (weeks) from date of remission status to disease relapse.
Time Frame: Throughout study, after each cycle for the first two cycles, then after every second cycle
Population: Remission duration was reported among participants who reported response
Measure: Mean (95% Confidence Interval); unit: Weeks
Arm/Group | Arm A, Step 1 | Arm A, Step 2 | Arm A, Step 3 | Arm A, Step 4 | Arm B, Steps 1-6 | Arm B, Step 7 | Arm B, Step 8 | Arm B, Step 9
Number analyzed (Participants) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Weeks |  | 26.3 [NA to NA] — Only 1 patient analyzed | 20.6 [NA to NA] — Only 1 patient analyzed |  | 5.4 [NA to NA] — Only 1 patient analyzed | 30.3 [NA to NA] — Only 1 patient analyzed | 19.6 [NA to NA] — Only 1 patient analyzed | 3.0 [NA to NA] — Only 1 patient analyzed

9. Secondary Outcome: Belinostat Cmax
Description: Cmax: Arm A: at Cycle 1 Day 4, Cycle 1 Day 5 Arm B: Cycle 1 Day 1 and Cycle 1 Day 2
Time Frame: Samples taken in Cycle 1 only, prior to initial dose on days 4 and 5 and at end of infusion, 5, 15, and 30 min, and 1, 2, 3, 4, and 6 hours post infusion
Population: Results shown for dose level 1000 mg/m2/d
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A, Cycle 1 Day 4 | Arm A, Cycle 1 Day 5 | Arm B, Cycle 1 Day 1 and Day 2
Number analyzed (Participants) | 18 | 17 | 15
ng/mL | 38744 (22653) | 31952 (16319) | 9657 (18859)

10. Secondary Outcome: Belinostat AUC (Area Under Curve)
Time Frame: Cycle 1, prior to initial dose on days 4 and 5 and at end of infusion, 5, 15, and 30 min, and 1, 2, 3, 4, and 6 hours post infusion
Population: Results shown for dose level 1000 mg/m2/d
Measure: Mean (Standard Deviation); unit: ng*hrs/mL
Arm/Group | Arm A, Cycle 1 Day 4 | Arm A, Cycle 1 Day 5 | Arm B, Cycle 1 Day 1 and Day 2
Number analyzed (Participants) | 18 | 17 | 15
ng*hrs/mL | 21850 (10327) | 21322 (7516) | 172823 (280715)

11. Secondary Outcome: Elimination t½
Time Frame: Cycle 1, Samples taken in Cycle 1 only, prior to initial dose on days 4 and 5 and at end of infusion, 5, 15, and 30 min, and 1, 2, 3, 4, and 6 hours post infusion
Population: Results shown for dose level 1000 mg/m2/d
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Arm A, Cycle 1 Day 4 | Arm A, Cycle 1 Day 5 | Arm B, Cycle 1 Day 1 and Day 2
Number analyzed (Participants) | 18 | 17 | 15
Hours | 12.7 (12.2) | 13.1 (10.2) | 4.21 (2.66)

ADVERSE EVENTS:
Arm/Group | Arm A, Step 1 | Arm A, Step 2 | Arm A, Step 3 | Arm A, Step 4 | Arm B, Steps 1-6 | Arm B, Step 7 | Arm B, Step 8 | Arm B, Step 9
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 2/3 | 7/9 | 2/7 | 2/3 | 6/6 | 6/7
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 9/9 | 6/7 | 3/3 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A, Step 1 (N=3) | Arm A, Step 2 (N=3) | Arm A, Step 3 (N=3) | Arm A, Step 4 (N=9) | Arm B, Steps 1-6 (N=7) | Arm B, Step 7 (N=3) | Arm B, Step 8 (N=6) | Arm B, Step 9 (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 2 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Anal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Central line infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Clostridium bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterococcal bacteriaemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary mycosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A, Step 1 (N=3) | Arm A, Step 2 (N=3) | Arm A, Step 3 (N=3) | Arm A, Step 4 (N=9) | Arm B, Steps 1-6 (N=7) | Arm B, Step 7 (N=3) | Arm B, Step 8 (N=6) | Arm B, Step 9 (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 5 | 2 | 1 | 3 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile Bone Marrow Aplasia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spontaneous Hematoma (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 2 | 3 | 3 | 0 | 3 | 4
Thrombotic Microangiopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac Disorder (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conduction Disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial Ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Antithrombin Iii Deficiency (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Macular Degeneration (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retinal Haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Visual Impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitreous Detachment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Anal Fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aphthous Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2 | 4 | 2 | 3 | 5 | 7
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 2 | 7 | 3 | 3 | 5 | 4
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tongue Blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tongue Discolouration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3 | 2 | 5 | 2 | 2 | 5 | 5
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Catheter Site Erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter Site Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter Site Related Reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 2 | 0
Face Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 4 | 1
Feeling Cold (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
General Physical Health Deterioration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Generalised Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion Site Pain (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Injection Site Reaction (General disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Localised Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal Inflammation (General disorders) | 0 | 2 | 1 | 2 | 0 | 0 | 2 | 1
Nodule (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 1 | 8 | 2 | 1 | 3 | 4
Pyrexia (General disorders) | 0 | 2 | 1 | 6 | 2 | 2 | 1 | 5
Visceral Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacterial Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchopulmonary Aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Central Line Infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Clostridium Bacteriaemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium Difficilie Colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enteritis Infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterobacter Bacteriaemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterococcal Bacteriaemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enterocolitis Infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fungal Skin Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes Simplex (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral Fungal Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pseudomonas Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary Mycosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Puncture Site Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Soft Tissue Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Allergic Transfusion Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Postoperative thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Splenic Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Wound Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Blood Bilirubin Increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Blood Cholesterol Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood Creatinine Increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 3
Blood Potassium Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Body Temperature Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Central Venous Pressure Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram Qt Prolonged (Investigations) | 0 | 0 | 0 | 1 | 2 | 1 | 3 | 1
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 1
Heart Rate Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
International Normalised Ratio Increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Ph Urine Deacreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet Count Decreased (Investigations) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Troponin T (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight Decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Weight Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
White Blood Cell Count Decreased (Investigations) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 0 | 1 | 3 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 2 | 0 | 1 | 5 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 3 | 2
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Movement Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Sleep Disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urethral Pain (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Blistering (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Blood Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2
Denture Wearer (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 2 | 2
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 2 | 1 | 0 | 2 | 3
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less